CLINICAL TRIAL: NCT06536738
Title: Esophageal Fistula After Anterior Cervical Decompression and Fusion
Acronym: ACDF
Status: Completed | Type: Observational
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Hua Luo, Department of Orthopedic, Taizhou Hospital
Other Study IDs: K20230934; 2024KY531 (Other Grant/Funding Number: Zhejiang Medicine and Health Scientific Research Project)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Fistula
MeSH Terms: conditions — Esophageal Fistula | interventions — Esophagoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: esophageal repair — The surgery confirmed a secondary esophageal fistula following the anterior cervical surgery. The procedure involved trimming the esophageal tissue around the fistula and repairing the fistula.

SUMMARY:
This study aims to evaluate the incidence, risk factors, and preventive measures of esophageal fistula following anterior cervical decompression and fusion. By understanding the mechanisms and clinical manifestations of this complication, the study seeks to provide clinicians with better guidelines for treatment and improve postoperative outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and older. Diagnosed with a secondary esophageal fistula following anterior cervical decompression and fusion surgery.

Postoperative confirmation of the esophageal fistula via imaging studies or endoscopy.

Presence of clinical symptoms such as dysphagia, coughing, or signs of infection.

Patients or their legal representatives must provide informed consent.

Exclusion Criteria:

Preexisting esophageal diseases such as esophageal cancer, severe esophagitis, or congenital anomalies.

Other types of fistulas not related to the surgery. Severe comorbid conditions, including: Uncontrolled diabetes, severe cardiovascular diseases, immunosuppression, pregnant women.

Individuals unable or unwilling to comply with study protocols. Life expectancy of less than six months due to other underlying health conditions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients secondary esophageal fistula following anterior cervical decompression and fusion surgery.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The healing rate after the repair of an esophageal fistula | 2 month
  Successful repair of an esophageal fistula can result in a high healing rate, with many patients experiencing complete recovery. However, complications such as infection, poor blood supply to the repaired area, or underlying health conditions can affect the healing process. Close postoperative monitoring and appropriate care are crucial to ensure optimal healing and to address any potential complications promptly.

IPD SHARING:
Plan to Share IPD: No